CLINICAL TRIAL: NCT00976859
Title: Efficacy of a Two-session Treatment of Cognitive Restructuring and Imagery Modification (CRIM) to Reduce the Feeling of Being Contaminated (FBC) in Adult Survivors of Childhood Sexual Abuse
Brief Title: Efficacy of Cognitive Restructuring and Imagery Modification to Reduce the Feeling of Being Contaminated After Childhood Sexual Abuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Regina Steil, PhD, Goethe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDIEBESCHMUTZTHEITI
Record Dates: First submitted 2009-09-14; First posted 2009-09-15 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Sexual Abuse; Posttraumatic Stress Disorder
Keywords: childhood sexual abuse; CSA; posttraumatic stress disorder; PTSD, feeling of being polluted; mental pollution, mental contamination; feeling of being contaminated; sexual assault; disgust, shame
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Cognitive Restructuring

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Waitlist control group (No Intervention)
  Interventions: Behavioral: Waitlist control group
- Imagery Modification (Experimental): Via a internet research patients collect data on skin renewal which is discussed afterwards; in a guided imagery modification the patients imagines the process of skin renewal and the building of new skin cells
  Interventions: Behavioral: Imagery Modification

INTERVENTIONS:
Behavioral: Imagery Modification — Research via internet concerning the frequency of skin exchange and disputation of the collected information; in the guided imagery modification the therapist instructs the patient to imagine the feeling of being contaminated and the process of peeling off their former contaminated skin and the maturing of hundreds of new clean skin cells
  Other Names: Cognitive Restructuring and Imagery Modification; CRIM
  Arms: Imagery Modification
Behavioral: Waitlist control group — Patients in the wait list control group are treated after a waiting period of five weeks
  Arms: Waitlist control group

SUMMARY:
The purpose of this study is to determine whether a short term programme with internet research on the frequency of skin exchange and guided imagery modification is effective in the treatment of the feeling of being contaminated in female victims of childhood sexual abuse (CSA).

DETAILED DESCRIPTION:
In the first session the women who suffer from a feeling of being contaminated after childhood sexual abuse are interviewed with the Structured Clinical Interview for DSM-IV (SCID) to ensure the clinical diagnosis of posttraumatic stress disorder and exclude women who meet the exclusion criteria. They get questionnaires and protocol sheets to fill out until the intervention session after a week. Afterwards the women are randomly assigned to an intervention group or a waitlist control group. During the intervention session the women in the intervention group research via internet how many times their skin cells in different regions of their body have exchanged since the sexual abuse to get the information that their skin has changed hundreds and hundreds of times and has nothing in common with their skin in childhood or adolescence. This first part of the intervention is based on a component of the DBT-PTSD. Afterwards the therapist guides an imagery modification. The women imagine the feeling of being contaminated and then to peel off their former contaminated skin and the maturing of hundreds of new clean skin cells to process the rational information of the internet research emotionally. At the end of the intervention session patients get a tape with the guided imagery instruction and commit to listen to the tape daily to exercise the guided imagery modification until the third session after a week. In the last session the homework is discussed and information on posttraumatic stress disorder and psychotherapeutic treatments of posttraumatic stress disorder is offered.Women in the waitlist control group get the same treatment as the women in the intervention group after a period of five weeks.

ELIGIBILITY:
Inclusion Criteria:

* Sexual abuse in childhood or adolescence
* Feeling of being contaminated
* Clinical diagnosis of posttraumatic stress disorder concerning the trauma of sexual abuse in childhood or adolescence according to DSM-IV
* Informed consent

Exclusion Criteria:

* Currently in psychotherapy
* Life time clinical diagnosis of schizophrenia, schizoaffective disorder or bipolar disorder according to DSM-IV
* Body mass index < 16,5
* Endangerment of self or others
* Clinical diagnosis of alcohol or drug addiction according to DSM-IV
* Mental retardation

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Intensity of the feeling of being contaminated (0-100: "not at all" till "extremely") | pre treatment, post treatment, follow up
Vividness of the feeling of being contaminated (0-100: "not at all" till "extremely") | pre treatment, post treatment, follow up
Distress associated to the feeling of being contaminated (0-100: "not at all" till "extremely") | pre treatment, post treatment, follow up

SECONDARY OUTCOMES:
Posttraumatic Diagnostic Scale | pre treatment, post treatment, follow up
Clinician-administered PTSD Scale | pre treatment, follow up
Rosenberg Self-esteem scale | pre treatment, post treatment, follow up
Beck Depression Inventory (BDI-II) | pre treatment, post treatment, follow up

CONTACTS AND LOCATIONS:
Overall Officials: Regina Steil, PhD, Principal Investigator — Department of Clinical Psychology and Psychotherapy of the Johann Wolfgang Goethe University of Frankfurt
Locations (1):
- Department of Clinical Psychology and Psychotherapy of the Johann Wolfgang Goethe University, Frankfurt am Main, Hesse, Germany

REFERENCES:
- See also: Related Info — http://www.studie.uni-frankfurt.de